CLINICAL TRIAL: NCT04241393
Title: An Open-label Trial to Evaluate the Absorption, Metabolism, and Excretion of a Single Dose of [14C]-Tavapadon in Healthy Adult Male Subjects at Steady State
Brief Title: An Open-label Trial to Evaluate Mass Balance of Tavapadon at Steady State in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-HV-001
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Suspensions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tavapadon (Experimental)
  Interventions: Drug: Tavapadon tablet; Drug: Tavapadon [14C] suspension

INTERVENTIONS:
Drug: Tavapadon tablet — Participants will receive multiple dose titration of Tavapadon (0.25 mg once daily [QD] on Days 1 to 3, 0.5 mg QD on Days 4 to 6, 1.0 mg QD on Days 7 to 9, 1.5 mg QD on Days 10 to 12, and 2.5 mg QD on Days 13 to 15)
Drug: Tavapadon [14C] suspension — Following 15-Day multiple dose titration of Tavapadon, participants will receive a single oral dose of Tavapadon 2.5 mg containing approximately 100 μCi of [14C] Tavapadon on Day 16

SUMMARY:
The purpose of this trial is to determine the absorption, metabolism, and excretion (AME) of [14C] tavapadon.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, ages 18 to 55 years, inclusive, at the time of signing the informed consent form (ICF).
2. Body mass index (BMI) of 18.0 to 32.0 kg/m2 and a total body weight > 50 kg (110 lbs).
3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, Gilbert's syndrome] is not acceptable) at Screening or Check-in as assessed by the investigator (or designee).
4. Male subjects with a pregnant or a nonpregnant partner of childbearing potential must agree to use an acceptable or a highly effective method of contraception from signing of informed consent during the trial, and for 7 days following the last dose of study drug.
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.
7. Capable of consuming the standard diet.
8. History of a minimum of 1 bowel movement per day.

Exclusion Criteria:

- Medical History and Concurrent Diseases

1. Has a history of psychotic symptoms requiring treatment with an antipsychotic medication within the 12 months prior to signing ICF.
2. Subjects with epilepsy, or history of epilepsy, or conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), or who have increased risk of seizures as evidenced by history of electroencephalogram with epileptiform activity. Subjects with a history of febrile seizures and/or history of head trauma with loss of consciousness requiring hospitalization overnight will be excluded as well.
3. Subjects with a current history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological disease that, in the opinion of the investigator or medical monitor, could compromise either subject safety or the results of the trial.

   Medical conditions that are minor or well controlled may be considered acceptable if the condition does not expose the subject to an undue risk of a significant AE or interfere with the assessments of safety during the course of the trial. The medical monitor should be contacted in any instance where the investigator is uncertain regarding the stability of a subject's medical conditions(s) and the potential impact of the condition(s) on trial participation.
4. Any condition possibly affecting drug absorption including history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed; cholecystectomy and bariatric weight loss surgeries will not be allowed).
5. History of substance or alcohol-use disorder (excluding nicotine; Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria) within 2 years prior to signing the ICF.
6. History of regular alcohol consumption exceeding 14 drinks/week [1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor] within 6 months prior to signing ICF.
7. Use of tobacco- or nicotine-containing products within 3 months prior to Check-in.
8. Subjects who answer "yes" on the Columbia-Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Item 4 or Item 5 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan, or Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting the criteria for C-SSRS Item 4 or Item 5 occurred within the last 6 months, OR

   Subjects who answer "yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting the criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR

   Subjects who, in the opinion of the investigator, present a serious risk of suicide.
9. Subjects who have attempted suicide in the past.

   - Physical Examination and Clinical Laboratory Results
10. Positive hepatitis panel (hepatitis B surface antigen and hepatitis C virus antibody) and/or positive human immunodeficiency virus test (HIV-1 and HIV-2 antibody) at Screening.
11. Positive urine drug screen (with cotinine) or positive alcohol breathalyzer at Screening and Check-in. Subjects with a positive drug screen for illicit drugs or cotinine are excluded and may not be retested or rescreened. Subjects with a positive urine drug screen resulting from use of marijuana (any cannabinoids), prescription medications, over-the-counter medications, or products that, in the investigator's documented opinion, do not signal a clinical condition that would impact the safety of the subject or interpretation of the trial results may continue evaluation for the trial following consultation and explicit approval by the medical monitor.
12. Subjects with a 12-lead ECG demonstrating the following:

    • QT interval corrected for heart rate using Fridericia's formula >450 msec (average of 3 ECGs obtained at the Screening Visit).
13. Subjects with any of the following abnormalities in clinical laboratory tests at the Screening Visit, confirmed by a single repeat measurement, if deemed necessary, and at the discretion of the investigator:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2 × upper limit of normal (ULN)
    * Total bilirubin ≥1.5 × ULN.
14. Subjects with other abnormal laboratory test results, vital sign results, or ECG findings unless, based on the investigator's judgment, the findings are not medically significant and would not impact the safety of the subjects or the interpretation of the trial results. The medical monitor should be contacted to discuss individual cases, as needed.

    Tests with exclusionary results should be repeated to ensure reproducibility of the abnormality before excluding a subject based on criteria provided in the protocol. For ECGs, 3 consecutive recordings are required and if 2 of the 3 remain exclusionary, then the subject is not eligible for the trial.

    - Disallowed Prior and Concomitant Medications
15. Subjects taking other prohibited medication or who would be likely to require prohibited concomitant therapy during the trial.

    - Other
16. Subjects with difficulty swallowing.
17. Subjects who are known to be allergic or hypersensitive to the IMP or any of its components.
18. Subjects who are known to be allergic or hypersensitive to contents of the standard diet.
19. Subjects who have participated in any clinical trial involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known) prior to dosing.
20. Receipt of blood products within 2 months prior to Check-in.
21. Donation of blood from 56 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
22. Poor peripheral venous access.
23. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in.
24. Subjects who have participated in a radiolabeled drug trial where exposures are known to the investigator within the previous 4 months prior to admission to the clinic for this trial or participated in a radiolabeled drug trial where exposures are not known to the investigator within the previous 6 months prior to admission to the clinic for this trial. The total 12-month exposure from this trial and a maximum of 2 other previous radiolabeled trials within 4 to 12 months prior to this trial will be within the CFR recommended levels considered safe, per US Title 21 CFR 361.1: less than 5,000 mrem whole body annual exposure with consideration given to the half-lives of the previous radiolabeled trial drugs received.
25. Any subject who, in the opinion of the sponsor, investigator, or medical monitor, should not participate in the trial.
26. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the investigator.
27. Unwilling or unable to comply with the lifestyle modifications described in this protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2020-11-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of [14C]-Tavapadon and Metabolites: Area under the radioactivity time curve from zero to infinity (AUCinf) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon and Metabolites: Area under the radioactivity time curve from time 0 to last quantifiable concentration (AUClast) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon and Metabolites: Peak radioactivity Cmax) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon and Metabolites: Time to last measurable radioactivity (Tlast) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon and Metabolites: Time to maximum radioactivity (Tmax) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon and Metabolites: elimination half-life (t½) for Tavapadon and Metabolites (PF-06752844), in plasma and whole blood | Day 16 up to Day 28
Pharmacokinetics of Tavapadon: Apparent total body clearance (CL/F) for Tavapadon | Day 16 up to Day 28
Pharmacokinetics of Tavapadon: Apparent volume of distribution (Vz/F) for Tavapadon | Day 16 up to Day 28
Ratio of Plasma AUCinf for Tavapadon to whole blood total Radioactivity AUCinf | Day 16 up to Day 28
Ratio of Plasma AUCinf for Metabolites (PF-06752844) to whole blood total Radioactivity AUCinf | Day 16 up to Day 28
Ratio of plasma AUCinf for Metabolites (PF-06752844) to plasma AUCinf for Tavapadon | Day 16 up to Day 28
Ratio of whole blood AUCinf for Tavapadon (and metabolites, measured as total radioactivity) to plasma AUCinf for Tavapadon (and metabolites, measured as total radioactivity) | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Total radioactivity in urine at different intervals | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Cumulative radioactivity excreted in urine (Cumulative Aeu) | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Fraction of the dose administered excreted in urine (Feu) for total radioactivity at different intervals | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Cumulative fraction of the dose administered excreted in urine (Cumulative Feu) for total radioactivity in urine | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Amount eliminated in feces (Aef) for total radioactivity in feces at different intervals | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Cumulative amount excreted in feces (Cumulative Aef) for total radioactivity in feces | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Fraction of the dose administered excreted in feces (Fef) for total radioactivity in feces at different intervals | Day 16 up to Day 28
Pharmacokinetics of [14C]-Tavapadon: Cumulative Fraction of the dose administered excreted in feces (Cumulative Fef) for total radioactivity in feces | Day 16 up to Day 28

SECONDARY OUTCOMES:
Number of Subjects with reported Treatment Emergent Adverse Events (TEAEs) | Up to Day 28
Number of subjects with Clinically significant changes in Electrocardiogram measures (PR,RR,QT and QTcF) | Up to Day 28
Number of subjects with Clinically meaningful changes in Vital signs (Systolic and Diastolic blood pressures, heart rate, respiratory rate and body temperature) | Up to Day 28
Number of subjects with clinically significant changes in laboratory measures | Up to Day 28
Change from baseline of the Columbia-Suicide Severity Rating Scale (C-SSRS) | At Baseline and up to Day 28
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, Study Director — Cerevel Therapeutics, LLC
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States